CLINICAL TRIAL: NCT00693550
Title: Oral Metal Contact Allergy: A Cause of Oral Squamous Cell Carcinoma?
Brief Title: Contact Allergies to Dental Metal as a Possible Risk Factor for Oral Cancer
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: James A. Yiannias M.D., Mayo Clinic Cancer Center
Other Study IDs: 497-00; P30CA015083 (NIH); CDR0000589036 (Other: Mayo Clinic)
Record Dates: First submitted 2008-06-06; First posted 2008-06-09 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-06

CONDITIONS: Head and Neck Cancer
Keywords: lip and oral cavity squamous cell carcinoma; oropharyngeal squamous cell carcinoma
MeSH Terms: conditions — Head and Neck Neoplasms; Lymphoid Interstitial Pneumonia; Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Other: metal patch tests — Twenty - seven (27) metal patch tests will be applied to the patient's back and left in place for 3 days

SUMMARY:
RATIONALE: Gathering information about allergies to metals may help doctors learn whether having an allergy to metal used in dental work increases the risk of developing oral cancer.

PURPOSE: This clinical trial is studying contact allergies to dental metal as a possible risk factor for oral cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Identify the relationship between intraoral metal contact allergy and epithelial carcinogenesis in patients with newly or previously diagnosed intraoral squamous cell carcinoma.
* Compare the prevalence of metal contact allergy in these patients with control data from other existing study populations.

OUTLINE: This is a multicenter study.

* Participants undergo metal patch testing using 27 metals* commonly used in dental repairs that are part of the Mayo metal series. Metal patches are applied to the patient's back for 3 days and the back is read on days 3 and 5. Relevant patient data obtained from their medical and dental history, physical exam, laboratory values and treatment are documented.

NOTE: *Healthy volunteers (control) undergo metal patch testing using 8 metals most commonly positive for contact allergens.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Meets 1 of the following criteria:

  * Newly or previously diagnosed oral squamous cell carcinoma

    * Recruited from the otorhinolaryngology departments of Mayo Clinic Rochester and Mayo Clinic Arizona
  * Healthy volunteer (control)

    * No history of intraoral squamous cell carcinoma
    * Employed at Mayo Clinic Rochester or Mayo Clinic Arizona

PATIENT CHARACTERISTICS:

* No immunosuppression
* No other conditions that interfere with patch testing

PRIOR CONCURRENT THERAPY:

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: otorhinolaryngology departments of Mayo Clinic Rochester and Mayo Clinic Arizona
Sampling Method: Non-Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2000-08; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Relationship between intraoral metal contact allergy and epithelial carcinogenesis | one year
Prevalence of metal contact allergy comparison to study control data | one year

CONTACTS AND LOCATIONS:
Overall Officials: James A. Yiannias, MD, Study Chair — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States